CLINICAL TRIAL: NCT05278377
Title: Effectiveness of the Apprenti en Action School-based Culinary Program on 9-10-year-old Children's Food Literacy and Vegetable and Fruit Consumption
Brief Title: Effectiveness of the Apprenti en Action School-based Culinary Program on 9-10-year-old Children's Food Literacy
Status: Completed | Type: Observational
Sponsor: Universite de Moncton (Other)
Collaborators: New Brunswick Innovation Foundation (Other)
Responsible Party: Principal Investigator, Stephanie Ward, Assistant professor, Universite de Moncton
Other Study IDs: 2122-006
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Fruit and Vegetable Intake; Eating Behavior
Keywords: School; Food skills; Cooking skills; Food literacy; Culinary program; Cooking program; Nutrition knowledge
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Apprenti en Action (intervention group): "Apprenti en Action" consists of six, one-hour culinary workshops offered once a week during school hours.
  Interventions: Behavioral: "Apprenti en Action" program
- Control group: Students in the control group do not receive the "Apprenti en Action" program.

INTERVENTIONS:
Behavioral: "Apprenti en Action" program — The "Apprenti en Action" program aims to teach students how to read and follow recipes, prepare and cook various foods using various culinary techniques, and apply food safety practices. Students are also taught the basics of healthy food, nutrition, and cooking.
  Groups: Apprenti en Action (intervention group)

SUMMARY:
In New Brunswick, Canada, only 53% of Kindergarten to Grade 5 students reported eating five or more vegetables and fruits per day in 2016-2017. Low intakes of vegetables and fruits are a marker for poor nutrition, which may impair the growth and cognitive development of children and adolescents and may put them at risk of developing certain non-communicable diseases earlier in life. It has been suggested that increasing children's food literacy may be an effective way of promoting healthier diets, including increasing vegetable and fruit intake among students. Since children spend most of their waking hours at school, this may be a key setting for promoting food literacy and healthy eating behaviors. Previous studies have found that culinary interventions that include taste testing and nutrition education may improve students' food literacy and vegetable and fruit consumption. Therefore, this quasi-experimental study aimed to assess the effectiveness of a school-based culinary program titled "Apprenti en Action" on primary school children's food literacy, breakfast, and vegetable and fruit consumption. Specifically, data were collected among Grade 5 students from ten francophone elementary schools, five of which received the "Apprenti en Action" program and five who did not. The "Apprenti en Action" program consisted of six, one-hour culinary workshops given once a week, at school, during school hours. Data on students' food literacy, breakfast, vegetable, and fruit consumption were collected via online questionnaires before and after the program. In addition to collecting quantitative data, qualitative data were collected from program participants and their parents to assess their perceptions of "Apprenti en Action".

DETAILED DESCRIPTION:
This study used a quasi-experimental design. Quantitative data from Grade 5 students from five francophone elementary schools in the province of New Brunswick, Canada, who participated in the "Apprenti en Action" culinary program were compared to those of Grade 5 students from five other elementary schools who did not receive the program. "Apprenti en Action" consists of six, one-hour culinary workshops offered once a week during school hours. The program aims to teach students how to read and follow recipes, prepare and cook various foods using various culinary techniques, and apply food safety practices. Students are also taught the basics of healthy food, nutrition, and cooking.

A questionnaire was developed based on previously-validated questionnaires and it measured vegetable and fruit consumption, breakfast consumption, concepts of food literacy including food and cooking skills as well as nutrition knowledge. All students will complete this self-administered online questionnaire before and after the program. Multilevel regressions will be used to assess the effectiveness of the culinary class on students' food literacy, breakfast, vegetable, and fruit consumption. Additionally, focus groups with children who participated in the "Apprenti en Action" program and their parents will be invited to share their perceptions of the program and how/if it has impacted the children's food literacy and eating behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Be enrolled in a Grade 5 or mixed Grade 4 and 5 class

Exclusion Criteria:

* None

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants are Grade 5 students enrolled in one of the 10 recruited francophone elementary schools in the province of New Brunswick, Canada.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in vegetable and fruit consumption at the end of the program | Baseline and Endpoint (Week 6)
  Students' consumption of vegetables and fruits was measured using two questions from the provincial New Brunswick Student Wellness Survey (New Brunswick Student Wellness Survey, 2016). These questions asked how many vegetables and fruits they had eaten the day before the survey. This was measured using a scale from 0 (None), to 7 (7 or more).
Change from baseline in breakfast consumption at the end of the program | Baseline and Endpoint (Week 6)
  Students' breakfast consumption was assessed based on one question from the provincial New Brunswick Student Wellness Survey (New Brunswick Student Wellness Survey, 2016). Students were asked to report how often they ate breakfast during the last school week. This question was scored from 0 (none) to 7 (7 days of the week).
Change from baseline in cooking skills at the end of the program | Baseline and Endpoint (Week 6)
  Cooking skills include all skills needed to prepare and cook foods, including cooking methods and food preparation techniques, and were measured using 18 questions. Among the questions, one was assessed with a five-point, downwards Likert-type scale (e.g. "Rate your ability to make the different breakfast foods"), and 17 questions were multiple-choice questions (e.g. "How long does it take to cook hard- and soft-boiled eggs?"). All cooking skills included in the questionnaire were skills that children were expected to have practiced during the program. The questionnaire was based on three previously-validated tools (Skeaff et al. 2020, Dean et al. 2021, Lavelle et al. 2017). Specifically, these questions measured children's ability to prepare breakfast, to use various cooking methods, to use kitchen equipment, to apply food safety practices, and to use various food preparation techniques. In total, a score ranging from 0 to 83 points was possible for this outcome variable.
Change from baseline in nutrition knowledge at the end of the program | Baseline and Endpoint (Week 6)
  Nine multiple-choice questions were used to assess children's nutrition knowledge, including their understanding of a balanced plate and food safety. These questions were inspired by those used in Skeaff et al.'s (2020) validated questionnaire. In total, a score of 0 to 9 points was possible for this outcome variable.
Change from baseline in food skills at the end of the program | Baseline and Endpoint (Week 6)
  Food skills represent the knowledge and skills required to choose and prepare food according to available resources and to cook balanced meals. They include meal planning, following a recipe, using leftovers, making and following a grocery list, reading nutrition labels, etc. Of the three questions used to measure food skills, two questions were multiple-choice questions (e.g. "The above picture is of French toast. What are three ingredients you need for French toast?") and one was a five-point downwards Likert-type scale ("From this list, indicate how good you are at performing these actions."). These questions were based on previously-validated questionnaires (Skeaff et al. 2020, Lavelle et al. 2017). In total, a score of 0 to 53 points was possible for this outcome variable.

SECONDARY OUTCOMES:
Student perception of the program | One week after the end of the program (Week 7)
  Students' perception of the program will be measured via virtual semi-structured focus groups. Two 40-45 minute sessions with 8-10 students per group are anticipated. Students will be asked to share their perception of the program's impact on their knowledge, skills, appreciation for healthy foods, and self-efficacy, as well as the strengths, weaknesses, and perceived relevancy of the program.
Parent perception of the program | One week after the end of the program (Week 7)
  Students' parents' perception of the program will be measured via virtual semi-structured focus groups. Two 40-45 minute sessions with 8-10 parents per group are anticipated. Parents will be asked to share their perception of the program's impact on their children's knowledge, skills, appreciation for healthy foods, and self-efficacy, as well as the strengths, weaknesses, and perceived relevancy of the program.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A Ward, PhD, RD, Principal Investigator — Universite de Moncton
Locations (1):
- Universite de Moncton, Moncton, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available to researchers upon reasonable request made to the principal investigator.

REFERENCES:
- [Background] Lavelle F, McGowan L, Hollywood L, Surgenor D, McCloat A, Mooney E, Caraher M, Raats M, Dean M. The development and validation of measures to assess cooking skills and food skills. Int J Behav Nutr Phys Act. 2017 Sep 2;14(1):118. doi: 10.1186/s12966-017-0575-y. PMID 28865452
- [Background] Dean M, Issartel J, Benson T, McCloat A, Mooney E, McKernan C, Dunne L, Brennan SF, Moore SE, McCarthy D, Woodside JV, Lavelle F. CooC11 and CooC7: the development and validation of age appropriate children's perceived cooking competence measures. Int J Behav Nutr Phys Act. 2021 Jan 30;18(1):20. doi: 10.1186/s12966-021-01089-9. PMID 33516243
- [Background] Miller LM, Cassady DL. The effects of nutrition knowledge on food label use. A review of the literature. Appetite. 2015 Sep;92:207-16. doi: 10.1016/j.appet.2015.05.029. Epub 2015 May 27. PMID 26025086
- [Background] Brown, J. (2019). Nutrition through the life cycle (7e ed.). Cengage Learning.
- [Background] Conseil de la santé du Nouveau-Brunswick. (2017). Sondage sur le mieux-être des élèves du Nouveau-Brunswick au niveau primaire de la maternelle à la 5e année (2016-2017) (p. 19). https://csnb.ca/sites/default/files/publications-attachments/sondage-mieux-etre-des-eleves-au-primaire-2016-2017-fr.pdf
- [Background] Dudley DA, Cotton WG, Peralta LR. Teaching approaches and strategies that promote healthy eating in primary school children: a systematic review and meta-analysis. Int J Behav Nutr Phys Act. 2015 Feb 25;12:28. doi: 10.1186/s12966-015-0182-8. PMID 25889098
- [Background] Evans CE, Christian MS, Cleghorn CL, Greenwood DC, Cade JE. Systematic review and meta-analysis of school-based interventions to improve daily fruit and vegetable intake in children aged 5 to 12 y. Am J Clin Nutr. 2012 Oct;96(4):889-901. doi: 10.3945/ajcn.111.030270. Epub 2012 Sep 5. PMID 22952187
- [Background] Skeaff, S., Govan, A., & Skeaff, M. (2020). A Practical Kitchen-Based Validation of the Food Skills Section of a Food Literacy Questionnaire for 9-10 Year Old Children.
- [Background] Maynard M, Gunnell D, Ness AR, Abraham L, Bates CJ, Blane D. What influences diet in early old age? Prospective and cross-sectional analyses of the Boyd Orr cohort. Eur J Public Health. 2006 Jun;16(3):316-24. doi: 10.1093/eurpub/cki167. Epub 2005 Sep 1. PMID 16141299
- [Background] Nathan N, Wolfenden L, Butler M, Bell AC, Wyse R, Campbell E, Milat AJ, Wiggers J. Vegetable and fruit breaks in Australian primary schools: prevalence, attitudes, barriers and implementation strategies. Health Educ Res. 2011 Aug;26(4):722-31. doi: 10.1093/her/cyr033. Epub 2011 May 13. PMID 21571836
- [Background] Neumark-Sztainer D, Wall M, Larson NI, Eisenberg ME, Loth K. Dieting and disordered eating behaviors from adolescence to young adulthood: findings from a 10-year longitudinal study. J Am Diet Assoc. 2011 Jul;111(7):1004-11. doi: 10.1016/j.jada.2011.04.012. PMID 21703378
- [Background] Wang Y, Bentley ME, Zhai F, Popkin BM. Tracking of dietary intake patterns of Chinese from childhood to adolescence over a six-year follow-up period. J Nutr. 2002 Mar;132(3):430-8. doi: 10.1093/jn/132.3.430. PMID 11880567
- [Background] Krebs-Smith SM, Heimendinger J, Patterson BH, Subar AF, Kessler R, Pivonka E. Psychosocial factors associated with fruit and vegetable consumption. Am J Health Promot. 1995 Nov-Dec;10(2):98-104. doi: 10.4278/0890-1171-10.2.98. PMID 10160052
- [Background] Karpouzis F, Lindberg R, Walsh A, Shah S, Abbott G, Lai J, Berner A, Ball K. Evaluating OzHarvest's primary-school Food Education and Sustainability Training (FEAST) program in 10-12-year-old children in Australia: protocol for a pragmatic cluster non-randomized controlled trial. BMC Public Health. 2021 May 22;21(1):967. doi: 10.1186/s12889-021-10302-0. PMID 34022839
- [Background] Harris G, Mason S. Are There Sensitive Periods for Food Acceptance in Infancy? Curr Nutr Rep. 2017;6(2):190-196. doi: 10.1007/s13668-017-0203-0. Epub 2017 Apr 29. PMID 28596932
- [Background] Baranowski T, Baranowski J, Cullen KW, Marsh T, Islam N, Zakeri I, Honess-Morreale L, deMoor C. Squire's Quest! Dietary outcome evaluation of a multimedia game. Am J Prev Med. 2003 Jan;24(1):52-61. doi: 10.1016/s0749-3797(02)00570-6. PMID 12554024